CLINICAL TRIAL: NCT03279094
Title: A Pilot Study of Pre-transplant Immunosuppressive Therapy for Haploidentical Transplants in Patients With Sickle Cell Disease
Brief Title: Haploidentical Transplantation With Pre-Transplant Immunosuppressive Therapy for Patients With Sickle Cell Disease
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17182
Record Dates: First submitted 2017-09-06; First posted 2017-09-12 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Hematopoietic stem cell transplantation; Haploidentical stem cell transplantation; Post-transplant Cytoxan
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Haploidentical stem cell transplantation (Experimental)
  Interventions: Biological: Hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: Hematopoietic stem cell transplantation — Haploidentical stem cell transplantation with pre-transplant immunosuppressive therapy

SUMMARY:
This is a study to evaluate the safety and toxicity of a treatment regimen consisting of 2 cycles of pre-transplant immunosuppressive therapy followed by myeloablative preparative regimen and allogeneic hematopoietic stem cell transplantation from a haploidentical donor in patients with sickle cell disease.

The overall goal of this study is to expand the donor pool for hematopoietic stem cell transplantation in sickle cell disease using haploidentical donors, and to develop a non-toxic, myeloablative regimen, with the goal of achieving a consistent donor chimerism utilizing pre-transplant immunosuppressive therapy.

DETAILED DESCRIPTION:
All patients will receive an haploidentical hematopoietic stem cell transplant with the following conditioning and GvHD prevention:

Pre-transplant immunosuppressive therapy:

2 cycles of Fludarabine and Dexamethasone x 5 days each cycle

Conditioning regimen:

rATG daily x 3 days, Fludarabine daily x 6 days and Busulfan daily x 4 days

GVHD prophylaxis:

Cyclophosphamide day +3 and +4, Tacrolimus and Mycophenolate mofetil

ELIGIBILITY:
Inclusion criteria

* Diagnosis: Patients with sickle cell anemia (Hgb SS or SB° Thalassemia) with baseline Hgb S more than 60%.
* Disease status:
* Significant neurologic event (stroke) or any neurological deficit lasting > 24 hours; or increased transcranial Doppler velocity (>200 m/s).
* History of one or more episodes of acute chest syndrome (ACS) in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. asthma therapy and/or hydroxyurea).
* History of one or more severe vaso-occlusive pain crises per year in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. a pain management plan and/or treatment with hydroxyurea).
* Recurrent priapism requiring medical therapy.
* Osteonecrosis of two or more joints despite the institution of supportive care measures.
* Prior treatment with regular RBC transfusion therapy, defined as receiving 8 or more transfusions per year for > 1 year to prevent vaso-occlusive clinical complications (i.e. pain, stroke, and acute chest syndrome)
* Echocardiograph finding of tricuspid valve regurgitation jet (TRJ) velocity ≥ 2.5 m/sec.
* Ages 1 to 30.
* Child Bearing Potential- Transplantation could be teratogenic and/or lethal to the developing fetus. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately.
* Informed Consent/Assent: All subjects must have the ability to understand and the willingness to sign a written informed consent.
* The recipient must have a related donor who is genotypically haploidentical on HLA-A, B, C and DRB1 loci.
* No HLA matched sibling or 10/10 matched unrelated donor is available.

Exclusion criteria:

* Any uncontrolled illness including ongoing or active bacterial, viral or fungal infection.
* Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to any in the pre- or post-transplant regimen.
* Pregnant women are excluded from this study.
* Patients with any active malignancy are ineligible for this study, other than non-melanoma skin cancers.
* Medical problem or neurologic/psychiatric dysfunction which would impair patient ability to be compliant with the medical regimen and to tolerate transplantation or would prolong hematologic recovery which in the opinion of the principal investigator would place the recipient at unacceptable risk.
* Prior autologous or allogeneic transplant.
* Fully HLA-matched related or unrelated donor is available to donate.
* Non-Compliance: Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2026-02-24 (Estimated); Study Completion 2026-02-24 (Estimated)

PRIMARY OUTCOMES:
Rate of unacceptable adverse events that are defined as any of the following events that occur from start of pre-transplant immunosuppressive therapy to the first 100 days post HCT: | 190 days
  * Rate of death of any causes
  * Rate of study discontinuation or early withdrawal
  * Rate of graft failure
    • Primary graft failure is defined as failure to achieve a neutrophil count of 0.5 x 109/L before day +42 or mixed chimerism with failure to achieve <30% Hgb S on electrophoresis after day +180. Secondary graft failure is defined as recovery followed by a sustained loss of initial graft.
  * Rate of grade 4 non-hematological toxicities per NCI CTCAE v4.03 that last more than 21 days

SECONDARY OUTCOMES:
Time to donor neutrophil engraftment | 24 months
  Day of Neutrophil Engraftment: The first of three consecutive days on which the ANC is ≥0.5x109/L
Time to donor platelets engraftment | 24 months
  Day of Platelet engraftment: The first documented day on which the platelet count is >20x109/L unsupported by platelet transfusions for 7 days
Rate of graft failure | 24 months
  Primary graft failure is defined as failure to achieve a neutrophil count of 0.5 x 109/L before day +42 or mixed chimerism with failure to achieve <30% Hgb S on electrophoresis after day +180. Secondary graft failure is defined as recovery followed by a sustained loss of initial graft.
Incidence of acute GvHD (grade II - IV) during the first 100 days after transplantation | 100 days after transplantation
Incidence of chronic GvHD | 24 months
Overall survival rate | 24 months
  • Overall survival: the time from start of PTIS to death, or last follow-up, whichever comes first.
Event-free survival rate | 24 months
  • Event-free survival: the time from start of PTIS to death, the unacceptable events, or last follow-up, whichever comes first.
Disease free survival rate | 24 months
  • Disease free survival: the time from HCT to death, secondary graft failure, or last follow-up, whichever comes first.
Immune reconstitution at day 100, 180 and 365 | 24 months
  • Immune reconstitution: measurement of CD3, CD4, CD8, CD11b, CD14, CD56, CD20/19, FoxP3+ Treg, and memory subsets.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 from start of pre-transplant immunosuppressive therapy to 24 months post transplant | 24 months post-transplant
Percent of donor chimerism at 12 and 24 months after HCT | 12 and 24 months after HCT
Change From Baseline in Pain Scores using Numerical Rating Scale or Faces Pain Rating Scale at 100 days, 6 months and 12 months post-transplant | 100 days, 6 months and 12 months post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Anna B. Pawlowska, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States